CLINICAL TRIAL: NCT04967287
Title: MyopiaX Treatment for the Reduction of Myopia Progression in Children and Adolescents: Safety and Efficacy Investigation
Acronym: MyopiaX-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dopavision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MyopiaX-1
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Myopia
Keywords: Digital treatment
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyopiaX (Experimental): MyopiaX treatment
  Interventions: Device: MyopiaX
- Myopia control spectacles (Active Comparator): Clinically validated treatment to control myopia
  Interventions: Device: Myopia control spectacles

INTERVENTIONS:
Device: MyopiaX — MyopiaX treatment twice a day
  Arms: MyopiaX
Device: Myopia control spectacles — To be used all as prescribed
  Arms: Myopia control spectacles

SUMMARY:
The purpose of this trial is to investigate the safety and efficacy of MyopiaX - a digital treatment intended to slow the progression of myopia in children and adolescents.

DETAILED DESCRIPTION:
The present study is a multicentric, randomized, controlled, single masked trial to investigate the signals of effect, the safety and tolerability of MyopiaX in slowing the progression of myopia.

The trial consists of 12 months treatment period. The first 6 months participants will be treated either with MyopiaX or with myopia control spectacles. During the second half of the trial, participants treated with MyopiaX will receive the myopia control spectacles in addition. 81 children and adolescent aged 6 - 12 years will be included in the trial. Eligible subjects will be randomly assigned in a 2:1 ratio to either the MyopiaX or the myopia control spectacles group.

ELIGIBILITY:
Inclusion Criteria:

* Myopic children (-0.75 to -5.0 D SER, least myopic meridian -0.50 D in each eye)
* At least VA 0.2 LogMAR in each eye
* Age: 6 - 12 years old
* Good tolerability of test session with VR system
* Binocular adequacy as tested with VR
* Ability to understand treatment and give valid assent

Exclusion Criteria:

* Concomitant or previous therapies for myopia
* Eye diseases/conditions:
* Anisometropia ≥ 1.5 D
* Astigmatism ≥ 3 D
* Ophthalmological comorbidities
* Optic nerve abnormalities
* Suspicion of syndromic or monogenetic myopia
* Systemic illnesses affecting eye health, eye growth, and/or refraction
* Any illnesses affecting dopamine function (e.g., sleep disorder)
* Medication affecting dopamine function, accommodation, pupil size, or having an impact on the ocular surface (such as allergy medications)
* Participation in other clinical studies
* Medical history (or family history) of photosensitive epilepsy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Change in axial length and in spherical equivalent refractive error | 6 months
  Change in axial length (mm) and in spherical equivalent refractive error )D)from baseline to month 6.

OTHER OUTCOMES:
Change in axial length and in spherical equivalent refractive error | 12 months
  Change in axial length (mm) and spherical equivalent refractive error (D) from month 6 to month 12
Retinal and choroidal imaging parameters | 12 months
  Retinal and choriodal parameters during the course of the trial
Device usability as measured with the user feedback questionnaire | 12 months
  Device usability as measured with the user feedback questionnaire at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ian Flitcroft, Prof., Study Chair — Centre for Eye Reserach Ireland, Technological University Dublin
Locations (10):
- Germany (5):
  - Suedblick GmbH, Augsburg
  - BeyondEye Clinic, Cologne
  - MVZ Makula-Netzhaut-Zentrum Breyer Kaymak Klabe, Düsseldorf
  - University Medical Center, Johannes Gutenberg- University, Mainz
  - University Eye Hospital Tübingen, Tübingen
- Erasmus University Medical Center, Rotterdam, Netherlands
- University of Minho, Braga, Portugal
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - University Complutense of Madrid, Madrid
- Moorfields Eye Hospital NHS Fundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loughman J, Lingham G, Kaymak H, Lorenz K, Polling JR, Beck A, Carracedo G, Dahlmann-Noor AH, Muller PL, Flitcroft I; MyopiaX-1 Study Group. MyopiaX-1 Safety and Efficacy of a Novel Approach to Slow Juvenile Myopia Progression: A Multicenter, Randomized, Controlled Trial. Ophthalmol Sci. 2025 Oct 10;6(1):100973. doi: 10.1016/j.xops.2025.100973. eCollection 2026 Jan. PMID 41438818